CLINICAL TRIAL: NCT02945891
Title: SElf-SAMpling in Cervical Cancer Screening. SESAM Study; a Key to Better Health. Clinical Validation of a Self-sampling Device in Patients With Cervical Cancer and Cervical Pre-invasive Neoplasia
Brief Title: SElf-SAMpling in Cervical Cancer Screening; SESAM Study
Acronym: SESAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Mari Nygård, Senior Medical Officer, Head of HPV-related Epiemiological Research Unit, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014/655; 5777899 (Other Grant/Funding Number: Cancer Society of Norway)
Record Dates: First submitted 2016-10-21; First posted 2016-10-26 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Cervical Cancer
Keywords: mass screening; coverage; self-sampling; clinical validity
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (Experimental): Each women recruited for the study belong to the study group. Intervention is performance of HPV testing on Evalyn®Brush and FloqSwab specimens compared to clinician-sampled specimen. Providing an urinary sample (Colli-PeeTM), blood, and a questionnaire data is optional.
  Interventions: Device: HPV testing of Evalyn®Brush, FloqSwab and Colli-Pee specimens

INTERVENTIONS:
Device: HPV testing of Evalyn®Brush, FloqSwab and Colli-Pee specimens — Each woman use the self-sampling devices in an advised order the day before they go to the hospital. There will be change of sampling order with every patient so that 50% of women will use Evalyn®Brush (Rovers Medical Devices, Oss, The Netherlands) first and 50% a FloqSwab (Coban Flock Technologies, Italy) first. In addition women are asked to provide a first void urine sample using a Colli-PeeTM (Novosanis, Belgium) on the same morning as the hospital visit. At the hospital clinician will take an additional specimen for which the performance of different self-sampling devices will be compared to.

SUMMARY:
Study aims to support development of evidence based health care in Norway through evaluating recently proposed technological improvements in cervical cancer control before their routine use. SESAM II study evaluates the accuracy of vaginal self-sampling for high risk human papillomavirus (hrHPV) testing compared with a physician-taken sample.

DETAILED DESCRIPTION:
Concept of collecting cervical cancer screening smear in home through self-sampling is new both for target population and medical professionals. Self-sampling increases screening attendance and could be an alternative to recruit more women to cervical cancer screening in Norway. As there are is an implementation ongoing to switch from cytology based screening to HPV based screening in Norway, a reliable self-sampling method for HPV testing should be available. Furthermore, detection of HPV from self-sampled specimen requires laboratory capacity and expertise to comply with quality assurance demands such as internal quality control, external quality assessment and quality improvement. National studies are crucial to obtain knowledge and build expertize among health care providers. This study aims to show non-inferior sensitivity of hrHPV testing on self-sampled vs. clinician-sampled specimens to detect high-grade cervical lesions and cancer (CIN2+). Additionally we will;

* Evaluate overall and hrHPV type specific concordance between self-taken and physician-taken samples.
* Evaluate participants views on feasibility and acceptability of self-sampling (questionnaire)
* Compare participants screening history with the questionnaire to evaluate the reason for not participating in the national screening program (if that is the case).
* Biobank biological material collected from self-sample, physician taken samples, blood and urine, for future analysis on HPV-related diseases and cancer.

Study participants will be recruited from the colposcopy referrals and cancer care units from three different hospitals. Patients with CIN 2 or CIN 3 lesions (n=200) will be recruited from Oslo University Hospital, Ullevål and Østfold Hospital Trust, while cancer patients (n=50) will be recruited from Radiumhospital.

ELIGIBILITY:
Inclusion Criteria:

* Women with histological verified CIN 2 or CIN 3
* Women with histological verified cervical cancer

Exclusion Criteria:

* Women with mild cervical lesions

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2014-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
High-risk HPV (hrHPV) testing on self-sampled specimens has non-inferior sensitivity for CIN 2+ compared to clinician-sampled specimens. | Sensitivity will be assessed through study completion, up to 36 months
  Relative sensitivity will be measured through histologically confirmed detection rates using clinician-sampled specimen as a reference.

SECONDARY OUTCOMES:
Overall and hrHPV specific concordance between self- and clinician-sampled specimens | Through study completion, an average of 6 months
  Agreement of hrHPV positivity rates between self-collected samples and physician-collected reference samples will be assessed by the kappa statistic.
Acceptability of feasibility of self-sampling | Through study completion, an average of 6 months
  We will evaluate the acceptability of different self-sampling devices based on the participants' views from a questionnaire.
Participants screening history and reasons for possible non-participation | Through study completion, an average of 6 months
  We will evaluate reasons for possible non-participation based on the participants' responses from a questionnaire and individual screening records at the Cancer Registry of Norway.

CONTACTS AND LOCATIONS:
Overall Officials: Giske Ursin, MD, Prof, Study Director — Oslo University Hospital, Cancer Registry of Norway
Locations (4):
- Norway (4):
  - Ostfold Hospital Trust, Fredrikstad
  - Oslo University Hospital, Molecular Pathology, Oslo
  - Oslo University Hospital, Ullevål, Oslo
  - Radiumhospital, Oslo

IPD SHARING:
Plan to Share IPD: No
We can't make individual participant data available due to restrictions set by the ethical approval and the informed consent. Our data contains several variables with personal health information, including age, dates, test results and diagnoses. Even without direct identifiers, it would be possible for a person to recognize herself from the dataset and that is strictly forbidden.

REFERENCES:
- [Derived] Leinonen MK, Schee K, Jonassen CM, Lie AK, Nystrand CF, Rangberg A, Furre IE, Johansson MJ, Trope A, Sjoborg KD, Castle PE, Nygard M. Safety and acceptability of human papillomavirus testing of self-collected specimens: A methodologic study of the impact of collection devices and HPV assays on sensitivity for cervical cancer and high-grade lesions. J Clin Virol. 2018 Feb-Mar;99-100:22-30. doi: 10.1016/j.jcv.2017.12.008. Epub 2017 Dec 21. PMID 29289814